CLINICAL TRIAL: NCT05544357
Title: Cardiovascular Adaptations to Resistance Exercise: Effects of Set Configuration on Normotensive and Hypertensive Postmenopausal Women
Brief Title: Cardiovascular Adaptations to Resistance Exercise: Effect of Set Configuration on Postmenopausal Women
Acronym: CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Eliseo Iglesias Soler, Principal Investigator, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PID2021-124277OB-I00
Record Dates: First submitted 2022-09-10; First posted 2022-09-16 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Postmenopausal; Hypertension
Keywords: resistance training; postmenopausal women; cardiovascular responses; cardiovascular adaptations
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resistance training with short set configuration performed by normotensive postmenopausal women (Experimental): Normotensive postmenopausal women performing resistance training protocol with the lowest cardiovascular stress identified in the first study of the project. It can be expected to be a short set configuration protocol
  Interventions: Other: Short set configuration resistance training
- Resistance training with short set configuration performed by hypertensive postmenopausal women (Experimental): Hypertensive postmenopausal women performing resistance training protocol with the lowest cardiovascular stress identified in the first study of the project. It can be expected to be a short set configuration protocol
  Interventions: Other: Short set configuration resistance training
- Resistance training with long set configuration performed by normotensive postmenopausal women (Experimental): Normotensive postmenopausal women performing resistance training protocol with the highest cardiovascular stress identified in the first study of the project. It can be expected to be a long set configuration protocol
  Interventions: Other: Long set configuration resistance training
- Resistance training with long set configuration performed by hypertensive postmenopausal women (Experimental): Hypertensive postmenopausal women performing resistance training protocol with the highest cardiovascular stress identified in the first study of the project. It can be expected to be a long set configuration protocol
  Interventions: Other: Long set configuration resistance training

INTERVENTIONS:
Other: Short set configuration resistance training — Resistance training protocol with the lowest cardiovascular stress identified in the first study of the project. It can be expected to be a short set configuration protocol
  Arms: Resistance training with short set configuration performed by hypertensive postmenopausal women; Resistance training with short set configuration performed by normotensive postmenopausal women
Other: Long set configuration resistance training — Resistance training protocol with the highest cardiovascular stress identified in the first study of the project. It can be expected to be a short set configuration protocol
  Arms: Resistance training with long set configuration performed by hypertensive postmenopausal women; Resistance training with long set configuration performed by normotensive postmenopausal women

SUMMARY:
The main purpose of this project is to analyze the effect of set configuration of resistance exercise on cardiovascular responses and adaptations of postmenopausal women. Additionally, since previous studies have shown that individual´s blood pressure level can influence on the impact of resistance training programs on cardiovascular changes, we aim to contrast acute and chronic changes to resistance training programs in normotensive and hypertensive postmenopausal women.

DETAILED DESCRIPTION:
Menopause causes hormonal changes that affect to acute and chronic physiological responses to exercise of postmenopausal women. In this regard, studies about the cardiovascular responses to resistance training in women are scarce, being particularly relevant to identify those load parameters that modulate these adaptations. Previous studies have identified that set configuration of muscular exercise influence on cardiovascular stress, albeit these results have been mainly obtained in healthy young male subjects.

The project is divided into two studies. The first one is devoted to contrast the acute effect of three resistance training sessions with the same volume, intensity, length a work-to-rest ratio, but differing in set configuration. Thus, a sample of 60 postmenopausal women (30 normotensive and 30 hypotensive) will be recruited in local sport facilities in order to carry out in a randomized order three experimental sessions and a control session. Before and after each session hemodynamic (systolic, diastolic and mean blood pressure), cardiac performance (heart rate, cardiac output, stroke volume among others), cardiac and vascular autonomic modulation (hear rate and blood pressure variability), baroreflex effectiveness (baroreflex sensitivity), neuromuscular fatigue, arterial stiffness and metabolic (lactate concentrations) responses and resting energy expenditure (oxygen consumption) will be evaluated. This first analysis will allow us to identify the two set configurations with the highest and the lowest cardiovascular stress respectively, being these exercise structures used in the second study, in which the effect of 12 weeks resistance training programs differing in set configuration will be contrasted. To do this, a sample of 40 postmenopausal women will be randomly assigned to a control group and to two resistance training programs (higher and lower set configuration respectively) which be carried out throughout 12 weeks with a frequency of 2 session per week. Training loads will be readjusted every four weeks. Before and after the training programs and after a 4 weeks follow-up period the following components will be evaluated: body composition by bioimpedance, muscular thickness by echography, neuromuscular performance (isokinetic torque-velocity and power-velocity relationship), resting metabolic rate by indirect calorimetry, foot bone mineral density, beat-to-beat blood pressure by photoplethysmography, cardiac performance by impedance cardiography , cardiac autonomic modulation by heart rate variability analysis, baroreflex sensitivity analysis, sympathetic vasomotor tone (blood pressure variability) and arterial stiffness. This project will provide useful information for optimizing the resistance exercise prescription for postmenopausal women by identifying exercise structures that potentially allow to preserve physiological adaptations and at the same time to blunt the acute cardiovascular stress.

ELIGIBILITY:
Inclusion Criteria:

* Five years since menopause
* Physically active (150-300 minutes a week of moderate physical activity or at least 75 minutes a week of vigorous physical activity)
* No more than 3 cardiovascular risk factors
* Asymptomatic and without cardiovascular (except hypertension), metabolic or renal disease
* Hypertensive women should be diagnosed with grade 1 hypertension that must be well controlled by one drug and with low or moderate cardiovascular risk.

Exclusion Criteria:

* Having grade 2 or 3 hypertension
* Participants with hypertension and taking more than one drug for controlling hypertension or by a drug that can interfere cardiovascular responses to exercise
* To be or have been receiving hormonal replacement therapy
* To show hypertensive response to exercise

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Baroreflex sensitivity | 25 minutes
  Simultaneous electrocardiogram and beat-to-beat blood pressure recordings obtained by a photoplethysmography sensor will be used for calculating baroreflex sensitivity by sequential methods. Units: mmHg/ms
Blood pressure | 25 minutes
  Systolic, diastolic and mean blood pressure will be obtained by a photoplethysmography sensor. Units: mmHg
Heart rate variability in time domain | 25 minutes
  Standard deviation of the normal-to-normal interval (SDNN) and root of the mean squared differences of successive NN intervals (RMSSD) will be obtained by analyzing inter-beat intervals from electrocardiogram recordings. Units: ms
Heart rate variability in frequency domain | 25 minutes
  Obtained from spectral analysis of electrocardiogram recordings. High (HF) and Low (LF) frequency bands power will be determined by Fast Fourier Transformation method. Units: ms2/Hz
Blood pressure variability | 25 minutes
  It will be calculated by spectral analysis of beat-to-beat blood pressure recordings obtained by a photoplethysmography sensor. Units: mmHg2/Hz
Resting metabolic rate | 60 minutes
  It will be obtained by measuring oxygen consumption at rest. Units: kcal/·day
Arterial stiffness | 15 minutes
  It will be assessed by finger-toe pulse wave velocity method. Units: m/s
Bone mineral density | 10 minutes
  It will be obtained by a Ultrasound Bone Densitometer. Units: g/cm

SECONDARY OUTCOMES:
Skeletal muscle mass | 10 minutes
  Estimated by Bioelectrical impedance analysis. Units: kg and percentage of body mass
Fat mass | 10 minutes
  Estimated by Bioelectrical impedance analysis. Units: kg and percentage of body mass
Body mass | 10 minutes
  Measured in kg
Body mass index | 2 minutes
  Measured in kg/m^2
Height | 10 minutes
  Measured in m
Muscle thickness | 20 minutes
  Measured with an ultrasound device. Units: mm
Torque-velocity relationship | 60 minutes
  Relationship between torque (N/m) and angular velocity (°/s). Obtained by performing maximum torque at specific velocities in an isokinetic dynamometer
Power-velocity relationship | 60 minutes
  Relationship betweenPower (W) and angular velocity (°/s). Obtained by performing maximum torque at specific velocities in an isokinetic dynamometer
Maximum isometric torque | 60 minutes
  Maximum torque recorded at fixed angular position. It will be measured with an isokinetic dynamometer. Units: N/m
Lipid profile to determine cardiovascular risk | 5 minutes
  * Total Cholesterol in mg/dL
  * High-Density Lipoprotein in mg/dL
  * Triglycerides in mg/dL
  * Calculated Low-Density Lipoprotein in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Eliseo Iglesias-Soler, PhD, Principal Investigator — University of A Coruna
Locations (1):
- Faculty of Sport Sciences and Physical Education, Bastiagueiro, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
After finishing the protocols (six months approximately) main data will be shared through European data repository Zenodo, in which University of A Coruna has created a community (https://zenodo.org/communities/udc/?page=1&size=20&size=20).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after finishing the whole project

REFERENCES:
- [Derived] Iglesias-Soler E, Farinas J, Rua-Alonso M, Rial-Vazquez J, Nine I, Revuelta-Lera B. Shorter Set Configurations Attenuate Performance Loss and Lactatemia During Resistance Training in Postmenopausal Women: A Randomized Crossover Trial (CARE Project). J Strength Cond Res. 2026 Feb 1;40(2):e180-e188. doi: 10.1519/JSC.0000000000005301. Epub 2025 Dec 5. PMID 41369549
- [Derived] Rial-Vazquez J, Rua-Alonso M, Enriquez-Gonzalez MG, Nine I, Rivera-Mejia SL, Revuelta-Lera B, Farinas J, Iglesias-Soler E. Cardiovascular adaptations to resistance training with different set configurations in postmenopausal women: a study protocol for a randomised controlled trial (CARE project). BMJ Open Sport Exerc Med. 2025 Nov 28;11(4):e003052. doi: 10.1136/bmjsem-2025-003052. eCollection 2025. PMID 41334240
- [Derived] Nine I, Padron-Cabo A, Carballeira E, Rial-Vazquez J, Rua-Alonso M, Farinas J, Giraldez-Garcia M, Iglesias-Soler E. Acute cardiovascular responses of postmenopausal women to resistance training sessions differing in set configuration: A study protocol for a crossover trial. PLoS One. 2024 Oct 14;19(10):e0311524. doi: 10.1371/journal.pone.0311524. eCollection 2024. PMID 39401188
- [Derived] Bohn L, Rial-Vazquez J, Nine I, Rua-Alonso M, Farinas J, Giraldez-Garcia MA, Mota J, Iglesias-Soler E. Arterial stiffness assessment by pulse wave velocity in postmenopausal women: comparison between noninvasive devices. Menopause. 2024 Aug 1;31(8):709-715. doi: 10.1097/GME.0000000000002383. Epub 2024 Jun 25. PMID 38916283